CLINICAL TRIAL: NCT03346083
Title: A Phase 1, Open-Label, Single-Dose, Non-Randomized Study to Evaluate Pharmacokinetics, Pharmacodynamics, and Safety of Betrixaban in Pediatric Patients
Brief Title: Study Evaluating Betrixaban in Pediatric Participants
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: After completion of Part 1 and prior to initiating Part 2, the Sponsor decided to cease developing betrixaban, prompting early study closure.
Sponsor: Alexion Pharmaceuticals, Inc. (Industry)
Collaborators: Portola Pharmaceuticals, LLC (a wholly owned subsidiary of Alexion Pharmaceuticals) (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-021; 2018-002562-40 (EudraCT Number)
Record Dates: First submitted 2017-11-07; First posted 2017-11-17 (Actual); Results first posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2023-04

CONDITIONS: VTE Prophylaxis
MeSH Terms: interventions — betrixaban

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cohort 1: Betrixaban 40 mg (Experimental): Participants received a single, oral dose of betrixaban at 40 mg in a fed state, and had 10 PK blood sampling time points.
  Interventions: Drug: Betrixaban
- Cohort 2: Betrixaban 80 mg (Experimental): Participants received a single, oral dose of betrixaban at 80 mg in a fed state, and had 5 PK sampling time points.
  Interventions: Drug: Betrixaban

INTERVENTIONS:
Drug: Betrixaban — Factor Xa inhibitor.
  Other Names: PRT054021

SUMMARY:
This trial was a Phase 1, open-label, multicenter study of the pharmacokinetics (PK), pharmacodynamics (PD), and safety of a single dose of betrixaban in pediatric participants at risk of venous thromboembolism (VTE).

DETAILED DESCRIPTION:
This study was to be conducted in 2 parts: Part 1 and Part 2. Part 1 (the initial opening of the study) was conducted in 21 adolescent participants (12 to < 18 years of age) who were assessed to be at risk for VTE. Participants in Part 1 received either 40 or 80 milligrams (mg) of study drug. The PK and PD data from Part 1 was to be used for dose determination for the next youngest age group using population PK and physiological-based PK modeling and simulation. Following analysis of Part 1 data, Part 2 of the study was to commence and enroll 12 participants 2 to < 12 years of age. However, after completion of Part 1 and prior to initiating Part 2, the Sponsor decided to cease developing betrixaban, prompting early study closure.

ELIGIBILITY:
Inclusion Criteria:

1. Pediatric participants in the following age categories: 12 to < 18 years of age and 2 to < 12 years of age. Part 1 of the study enrolled only adolescent participants 12 to < 18 years of age.
2. Pediatric participant who was assessed to be at risk for VTE but did not require immediate anticoagulant therapy, for example:

   1. Had previous thrombosis and completed a course of anti-coagulant therapy, and is considered to have a risk for recurrence of VTE, or
   2. Had any stable disease with a risk for arterial or venous thromboembolism, or
   3. Had any functional central venous access device in the upper or lower venous system.
3. Participant had normalized coagulation parameters (international normalized ratio or partial thromboplastin time, as appropriate) within 7 days of study drug administration.

Exclusion Criteria:

Participants who meet any one of the following exclusion criteria were excluded from the study:

1. Participant received any dose of anti-coagulant therapy within 7 days of Day 1.
2. Participant had active bleeding or had a comorbid disorder that placed the participant at high risk for bleeding.
3. Participant had a comorbid disorder that placed the participant at risk of death within 90 days of enrollment.
4. Participant had abnormal coagulation tests at baseline.
5. Participant had recent or planned invasive procedures, including lumbar puncture and removal of non-peripherally placed central lines during study.
6. Participant had hepatic disease associated with one or more of the following:

   * Transaminase levels ≥ 2.5 × upper limit of normal (ULN) or bilirubin ≥ 1.5 × ULN at baseline.
   * Coagulopathy leading to a clinically relevant bleeding risk, or hepatic transaminase level of > 2 × ULN or total bilirubin > 2 × ULN with direct bilirubin > 20% of the total.
   * Platelet count < 75 × 10^9/liter or hemoglobin < 10.0 mg/deciliter.
   * Hypertension.
7. Participant had known congenital or acquired bleeding diathesis.
8. Participant required concomitant therapy with a strong P-glycoprotein inhibitor.
9. Participant had previous history of any non-traumatic bleeding event that was life threatening or required medical attention.
10. Participant had been administered thrombolytic therapy, or had undergone thrombectomy, or insertion of a caval filter to treat prior VTE.
11. Participant had known inherited or acquired bleeding diathesis or coagulopathy.
12. Participant had abnormal QTcF interval on baseline electrocardiogram.
13. Participant received a dose of any antiplatelet medication (including aspirin) within 14 days before study drug dosing.
14. Participant had malabsorption disorders (for example, cystic fibrosis or short bowel syndrome).
15. Participant had an estimated glomerular filtration rate < 30 milliliters/minute.
16. Participant was unable or reluctant to cooperate with the study procedures.
17. Participant had hypersensitivity to other Factor Xa inhibitors, or the components of the dosage form.
18. Participant had participated in a study with an investigational drug or medical device within 30 days prior to administration of betrixaban.
19. Participant was female and of childbearing potential and was either pregnant or breastfeeding a child.
20. Participant was sexually active and was not using medically accepted contraceptive method (if applicable).

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 21 (Actual)
Dates: Start 2018-07-13 (Actual); Primary Completion 2019-10-08 (Actual); Study Completion 2019-10-08 (Actual)

CONTACTS AND LOCATIONS:
Locations (20):
- United States (5):
  - Children's Hospital Los Angeles, Los Angeles, California
  - ACTCA, Axis Clinical Trials, Los Angeles, California
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Tulane Medical Center, New Orleans, Louisiana
  - Rainbow Babies & Children's Hospital, Cleveland, Ohio
- Russia (6):
  - Children's Hospital of Tatarstan Republic, Kazan'
  - Federal State Institution, Kemerovo
  - Children's City Clinical Hospital, Moscow
  - Pirogov Russian National Research Medical University, Moscow
  - State Budgetary Institution, Nizhny Novgorod
  - Saint Petersburg State Pediatric Medical University, Saint Petersburg
- Ukraine (4):
  - Ivano-Frankivsk Regional Children Clinical Hospital, Ivano-Frankivsk
  - Odessa Regional Children Clinical Hospital, Odesa
  - Sumy Regional Children's Hospital, Sumy
  - Vinnytsia Regional Children's Clinical Hospital, Department of Anesthesiology and Intensive Care, Vinnitsa
- United Kingdom (5):
  - Birmingham Women's and Children's NHS Foundation Trust, Birmingham
  - Addenbrooke's Hospital, Cambridge
  - Children's Hospital for Wales, Cardiff
  - Glenfield Hospital, Leicester
  - Evelina London Children's Hospital, London

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: After a screening period of up to 30 days, eligible participants who had provided assent and for whom a parent or legal guardian had provided signed informed consent entered the hospital, clinical research unit, or Phase 1 unit on Day -1. Those who were already inpatients remained hospitalized.
Groups:
- Cohort 1: Betrixaban 40 mg: Participants received a single, oral dose of betrixaban at 40 milligrams (mg) in a fed state, and had 10 pharmacokinetic (PK) blood sampling time points.
Period: Overall Study
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Started | 3 | 18
Received At Least 1 Dose Of Study Drug | 3 | 18
Evaluated Through Day 7 Follow-up | 3 | 18
Completed | 3 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Enrolled population: all participants enrolled in Part 1 of the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg | Total
Number analyzed (Participants) | 3 | 18 | 21
Age, Customized [Count of Participants; unit: Participants]
  Age Categorical: In utero | 0 | 0 | 0
  Age Categorical: Preterm newborn - gestational age < 37 wk | 0 | 0 | 0
  Age Categorical: Newborns (0-27 days) | 0 | 0 | 0
  Age Categorical: Children (2-11 years) | 0 | 0 | 0
  Age Categorical: Adolescents (12-17 years) | 3 | 18 | 21
  Age Categorical: Adults (18-64 years) | 0 | 0 | 0
  Age Categorical: From 65 to 84 years | 0 | 0 | 0
  Age Categorical: 85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 9 | 11
  Male | 1 | 9 | 10
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 3 | 17 | 20
  Unknown or Not Reported | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 2 | 2
  White | 3 | 15 | 18
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United Kingdom | 0 | 1 | 1
  Ukraine | 0 | 2 | 2
  Russia | 3 | 11 | 14
  United States | 0 | 4 | 4

OUTCOME MEASURES:

1. Primary Outcome: Area Under The Plasma Concentration-Time Curve From 0 To Infinity (AUC(0-inf)) Of Betrixaban
Description: Following the Sponsor's decision to cease developing betrixaban, data for AUC(0-inf) were not collected.
Time Frame: Up to 6 days post dose
Population: After completion of Part 1 of the study and prior to initiating Part 2, the Sponsor decided to stop developing betrixaban and closed the study early. Therefore, data for this Outcome Measure were not collected.
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 0 | 0

2. Primary Outcome: Maximum Observed Plasma Concentration (Cmax) Of Betrixaban
Description: Data reported as "0.200" indicates that the data are below the lower limit of quantification. Note that the Measure of Central Tendency could not be determined for Cohort 1 or Cohort 2 due to the values that are below the lower limit of quantification.
Time Frame: Up to 6 days post dose
Population: The evaluable PK population included all participants who received the study drug and had sufficient blood samples through Day 3 to compute either Cmax or total AUC assessments with the extrapolated portion of the AUC(0-inf) less than 30%.
Measure: Geometric Mean (Full Range); unit: nanograms (ng)/milliliters (mL)
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 3 | 18
nanograms (ng)/milliliters (mL) | NA [0.200 to 2.57] — The Lower Limit and Upper Limit Cmax data are reported here as only individual participant data are available. | NA [0.200 to 48.5] — The Lower Limit and Upper Limit Cmax data are reported here as only individual participant data are available.

3. Secondary Outcome: AUC To The Last Measurable Concentration Above The Quantitation Limit (AUC(0-last)) Of Betrixaban
Description: Following the Sponsor's decision to cease developing betrixaban, data for AUC(0-last) were not collected.
Time Frame: Up to 6 days post dose
Population: as for outcome 1
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 0 | 0

4. Secondary Outcome: Terminal Plasma Half-life (t½) Of Betrixaban
Description: Following the Sponsor's decision to cease developing betrixaban, data for t½ were not collected.
Time Frame: Up to 6 days post dose
Population: as for outcome 1
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 0 | 0

5. Secondary Outcome: Time To Maximum Observed Plasma Concentration (Tmax) Of Betrixaban
Description: The Tmax that the highest (maximum) Cmax of betrixaban was observed per group up to Day 6 (120 hours) post dosing is reported.
Time Frame: Up to 6 days post dose
Population: as for outcome 2
Measure: Median (Full Range); unit: hours
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 3 | 18
hours | 2 [1 to 6] | 2 [1 to 12]

6. Secondary Outcome: Apparent Total Body Clearance Of Betrixaban From Plasma (CL)
Description: Following the Sponsor's decision to cease developing betrixaban, data for CL were not collected.
Time Frame: Up to 6 days post dose
Population: as for outcome 1
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 0 | 0

7. Secondary Outcome: Apparent Volume Of Distribution (Vd) Of Betrixaban
Description: Following the Sponsor's decision to cease developing betrixaban, data for Vd were not collected.
Time Frame: Up to 6 days post dose
Population: as for outcome 1
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 0 | 0

8. Secondary Outcome: Percent Change From Baseline In Thrombin Level At Day 6
Description: Following the Sponsor's decision to cease developing betrixaban, data for thrombin levels were not collected.
Time Frame: Baseline, Day 6
Population: as for outcome 1
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 0 | 0

9. Secondary Outcome: Count Of Participants With Treatment-related Adverse Events
Description: A treatment-related adverse event was any undesirable event or any untoward medical occurrence that occurs to a participant during the course of a study, or the protocol-defined time after study termination. An Investigator qualified in medicine made the determination of relationship to the investigational product for each adverse event (Unrelated, Unlikely Related, Possibly Related, or Probably Related). If the relationship between the adverse event and the investigational product was determined to be "possible" or "probable", the event was considered to be related to the investigational product for the purposes of expedited regulatory reporting. One participant experienced a mild study-drug-related headache that resolved in less than 2 hours. A summary of serious and all other non-serious adverse events, regardless of causality, is located in the Reported Adverse Events module.
Time Frame: Up to 7 days post dose
Population: Safety population: all participants enrolled in Part 1 of the study who received study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
Number analyzed (Participants) | 3 | 18
Participants | 0 | 1

ADVERSE EVENTS:
Time Frame: Up to 7 days post dose.
Arm/Group | Cohort 1: Betrixaban 40 mg | Cohort 2: Betrixaban 80 mg
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/18
Other Adverse Events (participants affected / at risk) | 0/3 | 5/18
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cohort 1: Betrixaban 40 mg (N=3) | Cohort 2: Betrixaban 80 mg (N=18)
Hypertension (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
Bradycardia (Cardiac disorders) | 0 (0) | 1 (1)
Headache (Nervous system disorders) | 0 (0) | 1 (1)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
After completion of Part 1 and prior to initiating Part 2, the Sponsor decided to cease developing betrixaban, prompting early study closure.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/83/NCT03346083/Prot_000.pdf
  • Statistical Analysis Plan (2020-06-02): https://cdn.clinicaltrials.gov/large-docs/83/NCT03346083/SAP_001.pdf